**PRINCIPAL INVESTIGATOR:** Alice P. Chen, M.D.

**STUDY TITLE:** A Phase II Trial in Which Patients With Metastatic Alveolar Soft Part Sarcoma Are Randomized to Either Sunitinib or Cediranib Monotherapy, With Cross-Over at Disease Progression

Progression

**STUDY SITE:** NIH Clinical Center

Cohort: Treatment

Consent Version: 6/3/2022

# WHO DO YOU CONTACT ABOUT THIS STUDY?

Alice P. Chen, MD, (240) 781-3320, chenali@mail.nih.gov Ashley Bruns, RN, (240) 858-3162, ashley.bruns@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers. Taking part in research at the NIH is your choice.

If the individual being enrolled is a minor then the term "you" refers to "you and/or your child" throughout the remainder of this document.

If the individual being asked to participate in this research study is not able to give consent for themselves, you, as the Legally Authorized Representative, will be their decision-maker and you are being asked to give permission for this person to be in this study. For the remainder of this document, the term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022


# WHY IS THIS STUDY BEING DONE?

The purpose of this study is to find out what effects, good and/or bad, the drugs cediranib and sunitinib have on you and your alveolar soft part sarcoma. This study will also help to find out how cediranib and sunitinib work in patients who have your type of cancer. The 2 drugs will not be given in combination during this study. You will receive one drug (either cediranib or sunitinib) until that drug is no longer working to control your cancer or you have too many side effects, and then the other drug will be given.

Cediranib is an experimental drug not yet approved by the Food and Drug Administration. Sunitinib has been approved for treating a certain type of kidney cancer and gastrointestinal cancer, but is considered experimental in the treatment of alveolar soft part sarcoma. Cediranib and sunitinib work by blocking the creation of new blood vessels. All solid tumors need new blood vessels to grow. We hope cediranib and sunitinib will stop tumor growth by preventing the growth of new blood vessels. So far, more than 800 patients have taken part in clinical trials of cediranib, including more than 40 patients with alveolar soft part sarcoma. More than 8,000 patients have received sunitinib, and at least 10 of these patients had alveolar soft part sarcoma. Some patients with alveolar soft part sarcoma treated with cediranib or sunitinib had tumors that either decreased in size or remained stable without growth for a prolonged period of time. Both cediranib and sunitinib are considered experimental drugs for your type of cancer.

#### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

Up to 70 patients with alveolar soft part sarcoma will take part in this study across several centers in the United States.

# DESCRIPTION OF RESEARCH STUDY

# What will happen if you take part in this research study?

After you are accepted for this study and you choose to take part, you will be "randomized" into one of the treatment groups (called "arms"). Randomization means that you are put into a group by chance. A computer program will place you in one of the treatment arms. Neither you nor your doctor can choose the treatment arm you will be in. This study is divided into two parts. During Part I, you will begin taking cediranib or sunitinib (depending on which arm you are in) by mouth once a day, every day. The treatment will be given in cycles. Each cycle is 28 days long. You will continue taking the study drug assigned to you (either cediranib or sunitinib) until that drug is no longer working to control your cancer, or you have too many side effects. After this happens, you will not get a study drug for 2 weeks before beginning Part II of the study. During Part II, you will receive the other study drug (either cediranib or sunitinib) that you did not take during Part I. However, if too many patients in a treatment arm have serious side effects or not enough patients have disease that responds, that treatment arm may be closed to new patients. If the other treatment arm is closed, you would not receive the other drug and your participation in the study would end after you complete Part I. Currently, the cediranib treatment arm for

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Page **2** of **20**IRB NUMBER: 11C0200

IRB APPROVAL DATE: 07/01/2022

1 - 5.85 -

patients with newly diagnosed ASPS is closed. No patients will enroll or cross over to this arm to receive cediranib.

Cediranib and sunitinib can be taken while you are an outpatient. You will take either cediranib or sunitinib during Part I and switch to the other drug during Part II. You are to swallow the tablets or capsules whole at about the same time each morning. Cediranib must be taken on an empty stomach, 1 hour before or 2 hours after meals. Sunitinib can be taken with or without food as you wish. You should write down the number of pills you take and the time you took them in the diary that your study team will give you. If you miss doses, please write this in your diary. If you remember your missed dose within 3 hours of the time you usually take a dose, you can take enough pills to make up for the missed dose; if not, do not make up the missed dose. The dose will be changed if you have any serious side effects. This will be determined by your study team.

# STANDARD PROCEDURES BEING DONE BECAUSE YOU ARE IN THIS STUDY; THESE MAY BE DONE MORE OFTEN BECAUSE YOU ARE IN THE STUDY:

- Clinic visit to ask how you are feeling and to evaluate you with a physical examination at the start of each cycle (every 4 weeks) (every 3 cycles for patients on study for 2 years or longer).
- Vital signs: You will need to have your vital signs (measurement of your temperature, breathing rate, and blood pressure) measured each time you are seen in the outpatient clinic. You will also need to have your blood pressure measured by a health care provider every 2 weeks for the first cycle of Part I and Part II. If you have high blood pressure and need medication to control it, the study doctor will tell you how often you will need to have your blood pressure checked during the study. We will also ask you to measure your own blood pressure at home each day for the entire study. If your blood pressure is ever more than 150/90, or if the diastolic pressure (the bottom number) increases by more than 20, you should call the research team. You should also call the research team if you experience any symptoms of high blood pressure, such as chest pain, shortness of breath, headache, blood in the urine, or double vision.
- **Blood tests:** Measurement of your white blood cells, red blood cells and platelets, and measurements of your blood sugar and electrolytes and of how your liver and kidneys work, will be done every 2 weeks for the first 2 cycles of Part I and Part II and then at the start of all other cycles (every 3 cycles for patients on study for 2 years or longer). Doing all of these blood tests will require 1-2 tablespoons (20-30 mL) of blood each time.
- Urine test: You will be asked to give a urine sample for testing at the start of each cycle (every 3 cycles for patients on study for 2 years or longer), or more often if your results have been abnormal. Depending on the results, you may be asked to collect your urine for 24 hours for further testing.
- **Pregnancy tests** in women who are able to become pregnant before you start cediranib or sunitinib and before you start Part II.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 Page **3** of **20** IRB NUMBER: 11C0200 IRB APPROVAL DATE:

- **EKGs** (a recording of the heart's electrical activity) to check your heart will be done before you start cediranib or sunitinib, before you start Part II, and at the start of each cycle (every 3 cycles for patients on study for 2 years or longer) to check for signs of possible damage to your heart.
- Echocardiogram to check your heart will be done before you start cediranib or sunitinib, before you start Part II, and at other times if needed to check for signs of possible damage to your heart. If abnormal, a repeat echocardiogram will be done every 2 cycles.
- CT scans (a computerized x-ray examination) or other imaging tests such as ultrasound (an examination using sound waves) or MRI (an examination using magnetic field and radio waves) that detect your tumor will be done every 2 cycles. PET scans (a scan that detects a small amount of radioactive substance that has been injected through a vein) will also be done at the start of the study and may be repeated. This is done so that any benefit of the drug can be seen, and so that if your cancer is not responding to the drug, the study team can tell you and help you move to a different treatment program (discussed further below).
- Magnetic resonance imaging (MRI) may be performed at the PI's discretion (instead of CT scans) prior to start of study treatment and then after every 2 cycles (about every 2 months) to measure your tumors.

MRI uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your body for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. We will place soft padding or a coil around your body segment being scanned. You will be in the scanner about 60 minutes. You may be asked to lie still for up to 60 minutes at a time. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at anytime. During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (IV) catheter. It will be done for both research and medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

# TESTS AND PROCEDURES THAT ARE EITHER BEING TESTED IN THIS STUDY OR BEING DONE TO SEE HOW THE DRUG IS AFFECTING YOUR BODY:

• Measurement of cediranib in your blood: We will collect multiple blood samples throughout the study to measure the amount of cediranib in your blood and to help us find out how the body handles cediranib. Please see the study chart for more details. The total blood for all these tests will be about 1~2 tablespoons.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# WHEN YOU ARE FINISHED TAKING STUDY DRUGS

You can take part in this study until either you or your study team decides that the study drugs are not helping you. If the first drug you are taking (either cediranib or sunitinib) is not helping you, you can move on to Part II of the study and receive the other drug if that treatment arm is open to new patients. Your taking part is voluntary, so you can stop taking cediranib or sunitinib at any time, but we ask that you speak to your study team before stopping the study drug.

Your study team will be watching you and your cancer during the study. If your cancer is clearly getting worse during Part II of the study, then your study team will stop the study treatment. At the end of the study, we will check with you or your local doctor for 30 days after you stop taking cediranib or sunitinib to see how you are doing. No more testing will be required.

# STUDY CHART

The treatment is given over 28-day periods of time called cycles. The 28-day treatment cycle will be repeated as long as you are not having serious side effects and your cancer is either steady or getting better. If the drug you receive during Part I of the study is no longer working to control your cancer or you have too many side effects, you can move on to Part II of the study and get the other drug if that treatment arm is open. Before you start Part II of the study there will be 2 weeks during which you get no study drug. This is called a "wash-out" period. You will also need to have certain tests repeated to make sure it is safe for you to start Part II of the study.

Each cycle is numbered. The chart below shows what will happen to you during Cycle 1 and future cycles. The left-hand column shows the day in the cycle and the right-hand column tells you what will happen on that day. This schedule lists what will happen to you after you sign the consent form and start the study. The cycle numbers will start at 1 again when you begin Part II of the study.

# Cycle 1 (Part I and Part II)

| Day | What to do and what will happen to you |
|---|---|
| Before | Check in at Outpatient Clinic |
| starting | Get routine blood and urine tests |
| study<br>treatment | • Have a history taken of how you feel and undergo a physical examination by a Health Care Provider (HCP) |
| | Imaging tests will be done |
| | EKG and echocardiogram will be done to check your heart |
| | Pregnancy test |

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# Cycle 1 and Future Cycles (Part I and Part II)

| Day | What to do and what will happen to you |
|---|---|
| Days 1-28 | Have a history taken of how you feel and undergo a physical examination by a Health Care Provider (HCP) at the start of each cycle |
| | • Get routine blood tests every 2 weeks for the first 2 cycles, then at the start of each cycle (every 3 cycles for patients on study for 2 years or longer) |
| | Urine sample for routine tests at the start of each cycle |
| | • Have your blood pressure checked by a health care provider every 2 weeks during cycle 1, then at the start of each cycle (every 3 cycles for patients on study for 2 years or longer). |
| | • Take cediranib or sunitinib, as given, once a day if you have no bad side effects and your cancer is not getting worse. Call the research nurse or your study doctor if you do not know what to do. |
| | Measure your blood pressure at home every day |
| | • Imaging tests will be done every 2 cycles to find out how your tumor is responding (every 3 cycles for patients on study for 2 years or longer) |
| | EKGs and echocardiograms will be done to check your heart |
| | • Blood samples to measure cediranib will be taken at the following time points before taking the drug: Before your first dose, on cycle 1 day 15, on cycle 2 day 1, on cycle 3 day 1, and on cycle 4 day 1. |

# STOPPING THERAPY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment (if this happens during Part I, you may still go on to Part II of the study, as long as the other treatment arm has not been closed)
- if you have side effects from the treatment that your doctor thinks are too severe (if this happens during Part I, you may still go on to Part II of the study, as long as the other treatment arm has not been closed)
- if new information shows that another treatment would be better for you

In this case, you will be told the reason why cediranib or sunitinib is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200


If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to the Cancer Therapy Evaluation Program (CTEP) at the National Cancer Institute (NCI) or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases **cannot** be recalled and destroyed.

# RISKS OR DISCOMFORTS OF PARTICIPATION

What side effects or risks can you expect from being in the study?

If you choose to take part in this study, there is a risk that the study drugs may not be as good as the usual approach for your cancer or condition at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The study drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study drug(s)/study approach.

Here are important things to know about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it hard for you to have children.
- Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

• If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

IRB APPROVAL DATE: 07/01/2022

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200


- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

• One patient on this study experienced bleeding in his brain around his cancer. The study drug may have contributed to the bleeding risk. This condition can keep oxygen from reaching the brain and cause brain damage or death.

Studies have shown high blood pressure to be one common side effect of cediranib and sunitinib. Your blood pressure will be closely watched while you are taking cediranib or sunitinib. This will include having your blood pressure measured every 2 weeks by a health care provider for the first cycle and you checking your blood pressure at home once a day for the entire study. If you have high blood pressure while taking cediranib or sunitinib, your study doctor may recommend follow-up with your primary care physician and/or starting or increasing medication to lower blood pressure.

We do not know if cediranib and sunitinib will have any effect on the bone growth of patients who have not finished growing. Please talk to your doctor or the research team about how this might affect the growth of a young patient.

Grapefruit juice has been shown to affect how the body handles some drugs by blocking the activity of the body's cytochrome P450 (CYP450) system. CYP450 is important in breaking down substances in the body, including sunitinib and many other drugs. Therefore, please avoid grapefruit juice while taking cediranib or sunitinib. The herbal supplement St. John's wort can also affect blood levels of drugs such as sunitinib, and should be avoided. We do not know if taking cediranib or sunitinib will cause other drugs you may be taking to work differently.

It is very important that you talk to a member of the research team before beginning any new drugs, over-the-counter medications, vitamins, or alternative therapies.

Risks and side effects related to cediranib include:

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving cediranib (AZD2171), more than 20 and up to 100 may have:

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBE


- Diarrhea, nausea
- Tiredness
- Loss of appetite
- Changes in voice
- High blood pressure which may cause headaches, dizziness, blurred vision

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving cediranib (AZD2171), from 4 to 20 may have:

- Pain
- Constipation, vomiting
- Dry mouth
- Difficulty swallowing
- Sores in the mouth
- Infection
- Bruising, bleeding
- Weight loss
- Dehydration
- Muscle weakness
- Dizziness, headache
- Cough, shortness of breath, sore throat
- Redness, pain or peeling of palms and soles
- Blood clot which may cause swelling, pain, shortness of breath, confusion, or paralysis

#### RARE, AND SERIOUS

In 100 people receiving cediranib (AZD2171), 3 or fewer may have:

- Anemia, kidney problems which may cause tiredness, bruising, swelling, or may require dialysis
- Heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or hole in internal organs that may require surgery
- Liver damage which may cause yellowing of eyes and skin, swelling
- Non-healing surgical site
- Damage to the brain which may cause changes in thinking
- Brain damage which may cause headache, seizure, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Kidney damage which may require dialysis
- Blood clot in artery which may cause swelling, pain, shortness of breath or change of color in extremity

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200

IRB APPROVAL DATE: 07/01/2022


#### Risks and side effects related to sunitinib include:

# **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving sunitinib malate (SU011248 L-malate), more than 20 and up to 100 may have:

- Pain
- Constipation, diarrhea, heartburn, nausea, vomiting
- Sores in the mouth
- Tiredness
- Loss of appetite
- Changes in taste
- Sore throat
- Redness, pain or peeling of palms and soles

# OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving sunitinib malate (SU011248 L-malate), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Blurred vision with chance of blindness
- Bloating, passing gas
- Dry mouth, skin
- Chills, fever
- Swelling of arms, legs
- Flu-like symptoms including body aches
- Bruising, bleeding
- Weight loss
- Infection, especially when white blood cell count is low
- Dehydration
- Dizziness, headache
- Feeling of "pins and needles" in arms and legs
- Depression
- Difficulty sleeping
- Cough, shortness of breath
- Nose bleed
- Hair loss, rash, itching, skin changes
- Change in hair color
- High blood pressure which may cause headaches, dizziness, blurred vision

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200


# RARE, AND SERIOUS

In 100 people receiving sunitinib malate (SU011248 L-malate), 3 or fewer may have:

- Anemia, kidney problems which may cause tiredness, bruising, swelling, or may require dialysis
- Blood clot which may cause confusion, paralysis, seizures or swelling, pain, shortness
  of breath
- Damage to organs (heart, brain, others) which may cause shortness of breath, swelling of ankles, and tiredness, changes in thinking
- Heart failure, heart attack which may cause shortness of breath, swelling of ankles, and tiredness
- Pain and swelling of thyroid
- Visual loss
- Difficulty swallowing
- A tear or hole in or between internal organs which may cause drainage and may require surgery
- Swelling of the gallbladder
- Liver damage which may cause yellowing of eyes and skin, swelling
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Flesh-eating bacteria syndrome
- Non-healing surgical site
- Change in the heart rhythm
- Kidney damage which may require dialysis
- Damage to the jawbone which may cause loss of teeth
- Damage to muscle which may cause muscle pain, dark red urine
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible) which may cause infection, bleeding, may require transfusions
- Stroke
- Brain damage which may cause headache, seizure, blindness (also known as Reversible Posterior Leukoencephalopathy Syndrome)
- Sores on the skin
- Severe skin rash with blisters and peeling which can involve mouth and other parts of the body

#### **Reproductive Risks**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we do not know how cediranib or sunitinib would affect your baby or your unborn child. You should not become pregnant or father a baby while on this study and for 2 months after you stop taking the drug because the drugs in this study can affect an unborn baby. It is important you understand that you and your partner need to use 2 forms of effective birth control (examples

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


below) while on this study and for 2 months after the study. Check with your study doctor about what kind of birth control methods to use and how long to use them. Some methods might not be approved for use in this study. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

abstinence

• intrauterine device (IUD)

• tubal ligation

- vasectomy
- hormonal [birth control pills, injections, or implants]

For more information about risks and side effects, please ask your study team.

#### **Risks for MRI**

People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

# Risks for Gadolinium-Enhanced MRI

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives,

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain.

#### **Radiation Risks**

During your participation in this research study, you will be exposed to radiation from CT scans. The amount of radiation exposure you will receive from these procedures is equal to approximately 7.7 rem per year. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." This study will expose you to more radiation than you get from everyday background radiation. No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The CT scan that you get in this study will expose you to the roughly the same amount of radiation as 26 years' worth of background radiation. Being exposed to too much radiation can cause harmful side effects such as an increase in the risk of cancer. The risk depends on how much radiation you are exposed to. Please be aware that about 40 out of 100 people (40%) will get cancer during their lifetime, and 20 out of 100 (20%) will die from cancer. The risk of getting cancer from the radiation exposure in this study is 0.77 out of 100 (0.77%) and of getting a fatal cancer is 0.38 out of 100 (0.38%).

#### POTENTIAL BENEFITS OF PARTICIPATION

# Are there benefits to taking part in the study?

The aim of this study is to see if either cediranib or sunitinib will cause your tumors to shrink. We hope that you will get personal medical benefit from taking part in this study, but we cannot be certain. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drugs' effect on your cancer, we do not know if you will benefit from taking part in this

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200


study, although the knowledge gained from this study may help others in the future who have cancer.

### ALTERNATIVE APPROACHES OR TREATMENTS

# What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems, and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# RESEARCH SUBJECT'S RIGHTS

# What are the costs of taking part in this study?

While you are on study at the National Cancer Institute, we will pay for the medications and treatments associated with the study. We cannot, however, assume the cost of your overall medical care. Any studies done outside of the NCI may require you or your insurance company to cover the cost of the service.

The study agents, cediranib and sunitinib, will be provided free of charge while you are participating in this study. Even though it is unlikely, there is a possibility that at some point the supply of study agent may run out necessitating taking you off-study. If this would occur, other possible options are:

- You might be able to get the cediranib or sunitinib from the manufacturer or your pharmacy but you or your insurance company may have to pay for it.
- If there is no cediranib or sunitinib available at all, no one will be able to get more and the study would close.

If a problem with getting cediranib or sunitinib occurs, your study doctor will talk to you about these options. You will not be paid for taking part in this study.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

# WHAT HAPPENS IF YOU ARE INJURED BECAUSE YOU TOOK PART IN THIS STUDY?

It is important that you tell your study team Principal Investigator Dr. Alice Chen at (240) 781-3320 if you feel that you have been injured because of taking part in this study. You will get medical treatment if you are injured as a direct result of taking part in this study at the NIH.

# WHAT ARE YOUR RIGHTS IF YOU TAKE PART IN THIS STUDY?

Taking part in this study is your choice. You may choose either to take part or to not take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. You can still get your medical care from our institution if you are eligible and choose to participate in another trial.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

#### CONFLICT OF INTEREST

The NIH reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The NIH and the research team for this study are using drugs developed by AstraZeneca and Pfizer Inc. through a collaboration between your study team and the company. The company also provides financial support for this study.

#### USE OF SPECIMENS AND DATA FOR FUTURE RESEARCH

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

My specimens and data may be kept for use in research to learn about, prevent, or treat cancer or other health problems.

Yes

No

**Initials** 

# COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

The NCI Developmental Therapeutics Clinic will cover some or all of your travel expenses related to participation in this study. This may include direct payments or reimbursements for expenses related to transportation, lodging, and meals. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. We will give you a copy of this policy.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


# CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study sponsor, the NCI Cancer Treatment Evaluation Program, or their agent(s).
- Qualified representatives from AstraZeneca, the pharmaceutical company who produces cediranib, and Pfizer, the pharmaceutical company who produces sunitinib.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

# PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 06/03/2022 IRB NUMBER: 11C0200


The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

#### **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Alice P. Chen, <a href="mail.mih.gov">chenali@mail.nih.gov</a>, (240) 781-3320. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

# **CONSENT DOCUMENT**

Please keep a copy of this document in case you want to read it again.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| <b>Adult Research Participant:</b> I hat to discuss it and to ask questions. | | planation about this study and have beer articipate in this study. | n given the opportunity |
|---|---|---|---|
| Signature of Research Participant | | Print Name of Research Participant | Date |
| about this study and have been give<br>to make research decisions on behavior | ven the opportual of the adult e, the informat | r an Adult Unable to Consent: I have<br>unity to discuss it and to ask questions. I<br>participant unable to consent and have t<br>cion in the above consent was described<br>e study. | am legally authorized he authority to provide |
| Signature of LAR | | Print Name of LAR | Date |
| | - | ave read the explanation about this study. I give permission for my child to take | |
| Signature of Parent/Guardian | | Print Name of Parent/Guardian | Date |
| Signature of Parent/Guardian | | Print Name of Parent/Guardian | Date |
| · · | | a way that I understand, I have been gitions. I agree to take part in this study. | iven the opportunity to |
| Signature of Minor | | Print Name of Minor | Date |
| Investigator: | | | |
| Signature of Investigator | | Print Name of Investigator | Date |
| Witness to the oral short-form c | onsent proces | es only: | |
| PATIENT IDENTIFICATION | Consent to 1 | Participate in a Clinical Research Stu | dy |
| | NIH-2977 (4-1 | 7)<br>4: Protocol Consent (1)<br>06/03/2022 IRB NUMBER: | • |

 $CC\ pre\ rCR\ ICF\ template\ v.\ 05.05.2020$ 

| MEDICAL RECORD | CONSENT T | O PARTICIPAT | E IN AN NIH C | LINICAL RESEARC | CH STUE |
|---|---|---|---|---|---|
| Signature of Witness* | | Print Name o | f Witness | Date | |
| *NIH ADMINISTRATIVE INTERPRETER: | SECTION TO | O BE COMPL | ETED REGAI | RDING THE USE | OF AN |
| An interpreter, or other in the administration of informe also serve as the witness. | | | | | |
| An interpreter, or other in the administration of informed providing interpretive support | l consent but did | <u>l not</u> serve as a w | | | |

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

